CLINICAL TRIAL: NCT05642468
Title: An Open Label, Phase 2 Study to Evaluate the Effect of A3907 on Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics in Adults With Primary Sclerosing Cholangitis (PSC)
Brief Title: Safety and Tolerability of A3907 in Primary Sclerosing Cholangitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albireo, an Ipsen Company (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3907-002; 2022-500790-14-00 (EU CTIS Number)
Record Dates: First submitted 2022-11-23; First posted 2022-12-08 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: PSC; Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 10 mg (Arm 1) (Experimental): 10mg tablet A3907 administered orally once daily for 12 weeks.
  Interventions: Drug: Ritivixibat
- 30 mg (Arm 2) (Experimental): 30mg (3x10 mg tablets) A3907 administered orally once daily for 12 weeks.
  Interventions: Drug: Ritivixibat
- 30 mg BID (Arm 3) (Experimental): 30mg (3x10 mg tablets) A3907 administered orally Bi-daily for 12 weeks.
  Interventions: Drug: Ritivixibat
- 30 mg BID for CRS (Arm 4) (Experimental): 30mg (3x10 mg tablets) A3907 administered orally Bi-daily for 12 weeks.
  Interventions: Drug: Ritivixibat

INTERVENTIONS:
Drug: Ritivixibat — 10mg tablet A3907 administered orally

SUMMARY:
This study will test a drug called A3907 to see how safe and tolerated it is for treating people with Primary Sclerosing Cholangitis (PSC).

DETAILED DESCRIPTION:
This study will test a drug called A3907 to see how safe and tolerated it is for treating people with Primary Sclerosing Cholangitis (PSC). Detailed Description: The primary goal of this study in participants with PSC with and without a Clinically Relevant Stricture (CRS) who are treated with A3907 is to assess the safety and tolerability of A3907 following repeat doses. Secondary goals include evaluation of the pharmacokinetic properties of A3907 (the study of how the body interacts with A3907 for the entire duration of exposure) and changes in safety parameters via laboratory testing such as liver enzymes, bile acid levels and markers of bile acid synthesis

ELIGIBILITY:
Key inclusion criteria:

1. Adults between 18 and 75 years of age (inclusive)
2. Clinical diagnosis of large-duct PSC as evidenced by chronic cholestasis with evidence of more than 6 months duration with either a consistent magnetic resonance cholangiopancreatography (MRCP) or endoscopic retrograde cholangiopancreatography (ERCP) showing sclerosing cholangitis. and historical evidence of elevated alkaline phosphatase (ALP).
3. Willing to sign informed consent.
4. Women of childbearing potential (WOCBP) and males with female partners of childbearing potential must agree to use contraception. Women of nonchildbearing potential (WONCBP) have a confirmatory follicle-stimulating hormone [FSH] level ≥ 40 mIU/mL
5. Alkaline phosphatase Phosphatase (ALP) value > 1.5 × upper limit of normal (ULN) but ≤ 10 × ULNULN at Visit 1 (Screening Period). Before starting 12 weeks treatment variability of < 30% between ALP values at Visit 1 and Visit 2 must be confirmed. If variability is > 30 % a third ALP value may be obtained. If the third ALP value meets >1.5 × ULN but ≤ 10 × ULN the patient can start the 12-week treatment period.
6. Arms 1-3 Only: Total bilirubin < 1.5 × ULN (unless due to Gilberts Syndrome or hemolysis) and normal direct bilirubin.
7. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 × ULN
8. Serum bile acid level > ULN
9. Arms 1 - 3 Only: An MRCP or equivalent imaging modality performed within 6 months before the Screening Period that is consistent with PSC without a clinically relevant stricture.
10. Arm 4 Only: An MRCP or equivalent imaging modality performed within 6 months before the Screening. Period that is consistent with PSC with a clinically relevant stricture, or clinically relevant bile duct obstruction (see Inclusion # 12 for additional information).
11. Use of ursodeoxycholic acid (UDCA) with a total daily dose ≤ 23 mg/kg/day, or bile acid-binding resins are permitted, with a minimum of 3 months of stable treatment prior to the Screening Period, and expected to remain on a stable dose through the 12-week treatment period; or a minimum of 3 months off UDCA prior to the Screening Period if UDCA was recently discontinued.
12. If a patient has inflammatory bowel disease (IBD) with a minimum disease duration of 4 weeks, this diagnosis should be documented. Inflammatory bowel disease should be in clinical remission or mildly active according to Crohn's Disease Activity Index (CDAI), partial Mayo score for Crohn's Disease (CD) and ulcerative colitis (UC), respectively (i.e. patients with CDAI score < 220 and Mayo score < 5, respectively). Patients with IBD should have had a colonoscopy performed within one year prior to the Screening Period with results showing no evidence of dysplasia or cancer
13. Clinically stable for at least 3 months prior to the Screening Period.
14. Arm 4 Only: One stable clinically relevant biliary stricture of at least 4 weeks duration on contrast-enhanced MRI/MRCP with > 75% reduction of duct diameter in the common bile duct or hepatic duct without suspicion of cholangiocarcinoma (further established by imaging and stable CA 19-9 below ULN repeated twice over 1 month), or cholelithiasis. Subjects may have signs or symptoms of worsening obstructive cholestasis (increasing jaundice, nausea, anorexia, steatorrhea and worsening or new onset pruritus), deterioration of liver function (i.e. decreasing platelet count, increasing international normalized ratio [INR]) and/could be listed for liver transplantation due to their clinically relevant biliary stricture.
15. Arm 4 Only: MELD Score < 35

Key exclusion criteria:

1. Presence of documented secondary sclerosing cholangitis, small duct PSC, known or suspected overlapping clinical and histologic diagnosis of autoimmune hepatitis or other causes of chronic liver disease
2. Arm 1-3 Only: Biliary intervention within 3 months prior to study enrollment or planned.
3. Arm 4 Only: Planned Biliary intervention between the Screening Period and baseline.
4. Presence of alternative causes of chronic liver disease, including alcohol-associated liver disease, nonalcoholic steatohepatitis, primary biliary cholangitis, autoimmune hepatitis, or active hepatitis B or C.
5. IBD with uncontrolled moderate to severe activity and/or on treatment with any immunosuppressive, immunomodulator, or biologic agent for treatment of IBD (i.e. azathioprine, 6 mercaptopurine, tacrolimus, methotrexate, infliximab, adalimumab, golimumab, vedolizumab, ustekinumab, tofacitinib, ozanimod). Treatment with corticosteroids (including budesonide, budesonide MMX and beclomethasone) in the previous 4 weeks.
6. History of human immunodeficiency virus infection or any other known relevant infection (e.g. tuberculosis).
7. History of ileectomy, colostomy or colectomy.
8. History of malignancy, including hepatocellular carcinoma and cholangiocarcinoma within the past 10 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated.
9. Alpha-fetoprotein (AFP) > 20 ng/mL (at the Screening Visit) with 4-phase liver CT or MRI suggesting presence of liver cancer.
10. History of transplants, including liver transplantation, or currently on active transplantation list (Arms 1 3). Arm 4 may be on an active liver transplantation list.
11. Current or a history of hepatic decompensation events including, but not limited to ascites, encephalopathy, or history of esophageal variceal bleeding.
12. Known or suspected overlapping clinical and histologic diagnosis of autoimmune hepatitis.
13. Small duct PSC (evidence of PSC on historical liver histology, with normal bile ducts on cholangiography) without large duct PSC.
14. Liver cirrhosis as assessed by any of the following:

    1. historical liver histology.
    2. liver stiffness measurement, assessed by FibroScan (FibroScan value > 14.4 kPa), in addition to clinical assessment and biochemical markers at the discretion of the investigator.
    3. signs and symptoms of hepatic decompensation (including, but not limited to, jaundice, ascites, variceal haemorrhage, and/or hepatic encephalopathy).
15. History of bacterial cholangitis within 60 days prior to the Screening Period, or if the patient is on antibiotics for prophylaxis of recurrent cholangitis.
16. Females who are pregnant, lactating, or breast feeding.
17. History of alcohol or substance abuse in the previous 2 years. Patients must agree to refrain from illicit drug (including marijuana) and alcohol use during the study.
18. Hypersensitivity to investigational medicinal product (A3907) and its excipients.
19. Presence of any contraindication for undergoing MRCP (e.g. pacemaker).
20. Any other condition or abnormality which, in the opinion of the investigator (or designee), may compromise the safety of the patient or interfere with the patient participating in, or completing the study.
21. Administration of medications that slow gastrointestinal motility.
22. Treatment with rifampicin.
23. Exposure to oral drugs that are strong inhibitors or inducers of CYP3A4 enzymes (e.g. grapefruit juice, ritonavir, itraconazole, ketoconazole, troleandomycin, rifampin, St John's wort, etc.) within 14 days prior to the Screening Period, or 5 half-lives of the drug, whichever is longer.
24. Exposure to oral drugs that are substrates of CYP3A4 enzymes (e.g. codeine, ciclosporin [cyclosporin], diazepam, etc.) during the study.
25. Treatment with vitamin D or fibrates, unless patient is on a stable dose ≥ 6 months prior to baseline.
26. Exposure to an investigational drug, biologic agent, or medical device within 30 days prior to the Screening Period, or 5 half-lives of the study agent, whichever is longer.
27. Platelet count < 150 000/mm3
28. Albumin level < 3.0 g/dL
29. INR > 1.3 (the patient may be treated with vitamin K intravenously, and if INR is ≤ 1.3 at resampling, the patient may be enrolled).
30. Medical conditions that may cause non-hepatic increases in ALP (e.g. Paget's disease). A GGT or ALP isoenzymes should be obtained for confirmation of biliary origin;
31. Glomerular filtration rate [GFR] < 60 mL/min/1.73 m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Treatment related adverse events | From baseline through week 12
  Number of participants with treatment related adverse events as assessed by CTCAE v 5.0

SECONDARY OUTCOMES:
Maximum observed plasma concentration and Area under the Plasma Concentration versus Time Curve (AUC) of A3907 | From baseline through week 12
Change in serum and urine individual and total bile acid levels | From baseline through week 12
  Measurement to see change in serum and urine individual and total bile acid levels
Change in ALT, AST, gamma-glutamyltransferase (GGT), ALP and bilirubin levels | From baseline through week 12
  Measurement to see change in ALT, AST, gamma-glutamyltransferase (GGT), ALP and bilirubin levels
Change in serum C4 level | From baseline through week 12
  Measurement to see change in 7α-hydroxy-4-cholesten-3-one (C4) and fibroblast growth factor 19 (FGF-19)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (8):
- Hopital Saint Antoine, Paris, France
- Italy (3):
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - ASST di Monza - Azienda Ospedaliera San Gerardo, Monza
  - Azienda Ospedale Università Padova, Padua
- Poland (3):
  - Centrum Medyczne INTER-MED, Częstochowa
  - Uniwersyteckie Centrum Kliniczne im. Prof. Kornela Gibinskiego, Katowice
  - ID Clinic Arkadiusz Pisula, Mysłowice
- Hospital Clinic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers